CLINICAL TRIAL: NCT00004762
Title: Phase II Pilot Study of Cladribine (2-Chlorodeoxyadenosine; 2-CdA) for Early Stage Primary Sclerosing Cholangitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: Scripps Clinic (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Purpose: Treatment
Other Study IDs: 199/11707; SCRF-94304
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2001-12

CONDITIONS: Cholangitis, Sclerosing
Keywords: gastrointestinal disorders; primary sclerosing cholangitis; rare disease
MeSH Terms: conditions — Cholangitis, Sclerosing; Gastrointestinal Diseases; Rare Diseases | interventions — Cladribine

INTERVENTIONS:
Drug: cladribine

SUMMARY:
OBJECTIVES:

I. Evaluate the effects of cladribine (2-chlorodeoxyadenosine; 2-CdA) on biochemical, radiologic, and histologic parameters in patients with early stage primary sclerosing cholangitis.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE:

Patients are treated with subcutaneous injections of cladribine (2-chlorodeoxyadenosine; 2-CdA) for 5 consecutive days every month for 3 months.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

Stage I-III primary sclerosing cholangitis

Radiologically and pathologically documented

No concomitant liver disease, e.g.:

* Viral hepatitis
* Autoimmune hepatitis
* Primary biliary cirrhosis
* Cirrhosis
* Portal hypertension or associated complications
* Jaundice caused by dominant stricture

--Prior/Concurrent Therapy--

No concurrent immunosuppressives

--Patient Characteristics--

Hematopoietic:

* Absolute neutrophil count at least 2500/mm3
* Platelet count at least 100,000/mm3
* Hemoglobin at least 10 g/dL

Other:

* No active infection
* No fistula abscess
* No active inflammatory bowel disease
* Quiescent disease allowed, including: Chronic ulcerative colitis Crohn's disease
* No other significant immunologic disorder
* No active malignancy
* No active alcohol or drug abuse
* No pregnant or nursing women
* Effective contraception required of fertile patients

Endoscopic retrograde cholangiopancreatography within 36 months prior to registration

Liver biopsy within 12 months prior to registration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5
Dates: Start 1994-12

CONTACTS AND LOCATIONS:
Overall Officials: Paul J. Pockros, Study Chair — Scripps Clinic